CLINICAL TRIAL: NCT07113106
Title: A Phase 1/2a Multicenter Trial to Evaluate the Safety and Immunogenicity of the CD40.Pan.CoV Vaccine, Adjuvanted or Not, as a Booster in Adult Participants
Brief Title: Dose Escalation Trial of CD40.Pan.CoV Vaccine, Adjuvanted or Not, as a Booster in Adult Healthy Volunteers
Acronym: PANCOV
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Enno DC (Unknown); Unité Mixte de Service 54 Methods and Applied Research for Trials (UMS 54 MART) (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2024-516767-92-01; ANRS0640s LKV-PAN-01 (PANCOV) (Other: Inserm-ANRS MIE)
Record Dates: First submitted 2025-06-18; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Healthy Volunteers
Keywords: a phase 1/2a, dose-escalating; Adult healthy volunteers; CD40.Pan.CoV vaccine adjuvanted or not; COVID19 vaccine; Safety and immunogenicity evaluation
MeSH Terms: interventions — poly ICLC

STUDY DESIGN:
Intervention Model Description: Pahse I/IIa multicenter dose-escalation trial to evaluate the safety and immunogenicity of the CD40.Pan.CoV vaccine, adjuvanted or not, as a booster in adult participants
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): Injection of Low dose CD40.Pan.CoV vaccine non adjuvanted
  Interventions: Biological: CD40.Pan.CoV Low dose(0.25mg)
- Cohort 2 (Experimental): Injection of LD CD40.Pan.CoV vaccine adjuvanted
  Interventions: Biological: CD40.Pan.CoV Low dose (0,25mg) adjuvanted with Hiltonol®
- Cohort 3 (Experimental): Injectionin of High dose CD40.Pan.CoV vaccine non adjuvanted
  Interventions: Biological: CD40.Pan.CoV High dose (1mg)
- Cohort 4 (Experimental): Injection of HD CD40.Pan.CoV vaccine adjuvanted
  Interventions: Biological: CD40.Pan.CoV High dose (1mg) adjuvanted with Hiltonol®

INTERVENTIONS:
Biological: CD40.Pan.CoV Low dose(0.25mg) — SC Injection in deltoid of Low dose (LD; 0.25 mg) CD40.Pan.CoV vaccine non adjuvanted at Day 0.
  Arms: Cohort 1
Biological: CD40.Pan.CoV Low dose (0,25mg) adjuvanted with Hiltonol® — SC injection in deltoid of LD (0.25 mg) CD40.Pan.CoV vaccine Hiltonol® adjuvanted at Day 0.
  Arms: Cohort 2
Biological: CD40.Pan.CoV High dose (1mg) — SC injectionin deltoid of High dose (HD; 1mg) CD40.Pan.CoV vaccine non adjuvanted at Day 0.
  Arms: Cohort 3
Biological: CD40.Pan.CoV High dose (1mg) adjuvanted with Hiltonol® — SC injection in deltoid of HD (1mg) CD40.Pan.CoV vaccine Hiltonol® adjuvanted at Day 0.
  Arms: Cohort 4

SUMMARY:
The clinical trial is a phase1/2a, open-label, dose-escalating, multicentre trial evaluating the safety and immunogenicity of the CD40.Pan.CoV vaccine, adjuvanted or not, as a booster injection in adult participants in France. 48 participants divided into 4 cohorts will be included in the trial.

Primary objectives are the following:

* To determine the safety and reactogenicity of different doses (0.25 mg and 1 mg) of a booster of a CD40.Pan.CoV vaccine, adjuvanted or not, in healthy volunteers between Day 0 and Month1
* To determine the humoral immune response (neutralizing antibody titers) induced by different doses (0.25 mg and 1 mg) of a booster of a CD40.Pan.CoV vaccine, adjuvanted or not, at Month1 after administration

DETAILED DESCRIPTION:
The ongoing COVID-19 pandemic continues to present a challenge to global public health and the response to the pandemic has been complicated by the rapid evolution of the virus.

Even though vaccinations have reduced severe cases, the constant appearance of new variants has decreased the effectiveness of current vaccinations. The development of more effective vaccines is therefore becoming necessary.

Two main concerns leave open scientific and policy questions regarding the optimal use and further development of COVID-19 vaccines and represent public health challenges and preventing the morbidity/mortality related to SARS-CoV-2 (re) infections. First, the continuous appearance of SARS-CoV-2 variants causing virus escape from vaccine and/or natural infection, humoral responses and second the durability of vaccine-induced protective immunity from infection.

Although certain data are reassuring with the current vaccines - in particular the conservation of the T response against variants - it is clear that vaccines incorporating additional T-cell antigens, acting in synergy with antibodies, may prove beneficial in preventing both infection and serious diseases induced by SARS-CoV-2 variants and future coronaviruses, and would avoid the need for annual or bi-annual renewal of current vaccines.

From this perspective, the CD40.Pan.CoV will be assessed in this trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 and <65 years at the day of screening.
2. Able to understand and comply with planned trial procedures and willing to be available for all trial-required procedures, visits and calls for the duration of the trial.
3. Voluntarily signed written informed consent before performance of any trial-related screening procedures.
4. Being covered by the Health Insurance.
5. Agree to be registered in the French Health Ministry computerized file.
6. In healthy condition or with stable health status which is defined as an existing disease that has not required a significant change in treatment or hospitalization for worsening before enrolment, and for which neither a significant change in treatment or hospitalization for worsening is expected in the near future.
7. Subject who has received a primary series of vaccination and ≥ 1 booster(s) of COVID-19 mRNA vaccination(s) with the last boost at least 6 months prior to the inclusion in the trial (i.e. 2 doses of vaccine for subjects with a history of COVID-19 infection and 3 doses of vaccine for subjects with no history of COVID-19 infection).
8. Subject who has normal biological values:

   * ALT, AST, and alkaline phosphatase < 1.25 x ULN (Liver function)
   * Creatinine < 1.1 x ULN of the laboratory
   * Hemoglobin ≥ 11.0 g/dL for females and ≥ 13.0 g/dL for males
   * Platelets = 125,000 to 550,000/mm3
   * White blood cell count = 3,300 to 12,000 cells/mm3
   * Total lymphocyte count ≥ 800 cells/mm3 Biological parameters outside of these values should be reviewed by the clinician who should specify the clinically significance. Results considered non-clinically significant by the clinician are accepted.
9. Virology assessment:

   * Negative Hepatitis B surface antigen (HBsAg)
   * Negative anti-Hepatitis C virus antibodies (anti-HCV), or negative HCV polymerase chain reaction (PCR) if the anti-HCV is positive.
   * Negative HIV antigen/antibody test
10. Normal urine test:

    * Negative urine glucose, and
    * Negative or trace urine protein, and
    * Negative or trace urine hemoglobin (if trace hemoglobin is present on dipstick, a microscopic urinalysis should show red blood cells levels within institutional normal range. Results considered non-clinically significant by the clinician will be accepted).
11. For women of childbearing potential: a negative Beta-HCG blood test measure during the screening visit, and a negative highly sensitive pregnancy urinary test the day of the vaccination visit AND use of a highly effective contraceptive method at least 4 weeks prior to vaccination and until at least 4 months after the vaccination.

    Highly effective contraception is defined as using any of the following methods:
    * Combined hormonal contraception with inhibition of ovulation (estrogen and progesterone containing)
    * Intrauterine device;
    * Intrauterine hormone releasing system;
    * Hormonal contraception (progesterone only);
    * Successful vasectomy in the male partner (considered successful if a participant reports that a male partner has (i) documentation of azoospermia by microscopy, or (ii) a vasectomy more than 2 years ago with no resultant pregnancy despite unprotected sexual activity post vasectomy);
    * Or not be of reproductive potential, such as having reached menopause (no menses for 1 year without an alternative medical cause) or having undergone hysterectomy, bilateral oophorectomy, or tubal ligation.

    For male participants: Willing to use an effective method of contraception with their partner (condoms) from the first day of IMP administration until 4 months after the administration. This also applies to sperm donation.
12. Willingness to undertake SARS-CoV-2 testing according to trial protocol, and receive SARS-CoV-2 test results.

Exclusion Criteria:

1. Acute febrile infection (body temperature ≥ 38.0°C) within the previous 72 hours and/or presenting symptoms suggestive of COVID-19 or SARS-CoV-2 infection within the previous 28 days or having been in contact with an infected individual for the last 14 days before the inclusion visit.
2. Immunosuppressive medications received within the last three months before IMP administration or within 6 months for chemotherapies. (Not excluded: [1] corticosteroid nasal spray; [2] topical corticosteroids for mild, uncomplicated dermatitis; or [3] a single course of oral/parenteral corticosteroids at doses < 2 mg/kg/day and length of therapy < 11 days with completion at least 30 days prior to enrolment). The scheduled use of these treatments up to 6 months after the injection also represents a contraindication.
3. Immunoglobulins and/or monoclonal antibodies within 90 days before IMP administration. The scheduled use of these treatments up to 6 months after the injection also represents a contraindication.
4. Blood products, including convalescent plasma, within 120 days before IMP administration. The scheduled use of these treatments up to 6 months after the injection also represents a contraindication.
5. Any medical condition that could impair the immune response: clinically significant medical condition (like cancer), clinical examination findings, clinically significant abnormal laboratory results, or past medical history with clinically significant implications for current health. A clinically significant condition or process includes but is not limited to:

   * A process that would affect the immune response;
   * A process that would require medication that affects the immune response;
   * Any contraindication to repeated injections or blood draws;
   * A condition that requires active medical intervention or monitoring to avert grave danger to the participant's health or well-being during the trial period;
   * A condition or process for which signs or symptoms could be confused with reactions to vaccine;
   * Any condition specifically listed among the exclusion criteria below.
6. Intent to participate in another trial of an investigational research agent within 4 weeks prior to the enrolment visit or until the end of follow-up.
7. Under tutorship, guardianship, or deprived of liberty by a juridical or administrative decision.
8. Pregnancy or breastfeeding that is currently ongoing, or positive pregnancy test at screening visit and the day of the vaccination.
9. History of severe adverse events following vaccine administration including anaphylactic reaction and associated symptoms such as rash, breathing problems, angioedema, and abdominal pain, or a history of allergic reaction that could be triggered by a component of the SARS-CoV-2 vaccine at the time of the vaccine injection (Not excluded: a participant who had a non-anaphylactic adverse reaction to pertussis vaccine as a child).
10. Any bleeding disorder considered as a contraindication to an intramuscular injection, previous phlebotomy, or receipt of anticoagulants.
11. A condition that requires active medical intervention or monitoring to avert grave danger to asthma other than mild, well-controlled asthma (symptoms of asthma severity as defined in the most recent National Asthma Education and Prevention Program (NAEPP) Expert Panel report). Exclude a subject who:

    * Uses a short-acting rescue inhaler (typically a beta 2 agonist) daily, or
    * Uses moderate/high dose inhaled corticosteroids, or
    * In the past year has either of the following: (i) Greater than 1 exacerbation of symptoms treated with oral/parenteral corticosteroids or (ii) Needed emergency care, urgent care, hospitalization, or intubation for asthma.
12. Hypertension:

    * If a person has been diagnosed with hypertension, exclude for blood pressure that is not well controlled (well-controlled blood pressure is defined as consistently ≤ 140 mm Hg systolic and ≤ 90 mm Hg diastolic, with or without medication, with only isolated, brief instances of higher readings, which must be ≤ 150 mm Hg systolic and ≤ 100 mm Hg diastolic). For these participants, blood pressure must be ≤ 140 mm Hg systolic and ≤ 90 mm Hg diastolic at enrolment
    * If a person has NOT been diagnosed with hypertension, exclude for systolic blood pressure ≥ 150 mm Hg at enrolment or diastolic blood pressure ≥ 100 mm Hg at enrolment (the measurement must be performed on a person who has been lying down for at least 5 minutes and repeated at the end of the consultation, if appropriated). Tension must be confirmed outside the clinical site to rule hypertension.
13. BMI ≥ 40 kg/m2; ≤ 18 kg/m2; or BMI ≥ 35 kg/m2 with 2 or more of the following: age > 45, current smoker, known hyperlipidemia, blood pressure is defined as consistently ≥ 140 mm Hg systolic and ≥ 90 mm Hg diastolic.
14. Malignancy (Not excluded: participant who has had malignancy excised surgically and who, in the investigator's estimation, has a reasonable assurance of sustained cure, or who is unlikely to experience recurrence of malignancy during the period of the trial).
15. Asplenia: any condition resulting in the absence of a functional spleen.
16. Seizure disorder: History of seizure(s) within the past three years. Also exclude if Participants have used medications to prevent or treat seizure(s) at any time within the past 3 years.
17. History of hereditary angioedema, acquired angioedema, or idiopathic angioedema.
18. History of myocarditis, pericarditis, cardiomyopathy, congestive heart failure with permanent sequelae, clinically significant arrhythmia (including arrhythmia requiring medication, treatment, or clinical follow-up).
19. History of autoimmune disease.
20. Any medical, occupational, or other condition that, in the judgment of the investigator, would interfere with or serve as a contraindication to protocol adherence, assessment of safety or reactogenicity, or a participant's ability to give informed consent.
21. Psychiatric condition that precludes compliance with the protocol. Specifically excluded are persons with psychoses within the past 3 years, ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years.
22. Any vaccination received within 30 days before IMP administration.
23. Allergy treatment with antigen injections within 30 days before IMP administration. The scheduled use of these treatments up to 6 months after the injection also represents a contraindication.
24. Other prohibited medications: Corticosteroids > 10 mg prednisone equivalent/day (not excluded: topical preparations), Immunomodulators (such as cytokines or interferons) and anti-tuberculosis drugs within 3 months before IMP administration. The scheduled use of these treatments up to 6 months after the injection also represents a contraindication.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-06-18 (Actual); Primary Completion 2026-06-25 (Estimated); Study Completion 2027-06-25 (Estimated)

PRIMARY OUTCOMES:
Safety primary outcome | From Day 0 (injection) to Month 1
  • Proportion of participants without any grade 3 or 4 solicited local/systemic or unsolicited AEs after the vaccine administration and considered to be related or possibly related to IMP administration
Immunogenicity primary outcome | from Day 0 (vaccine injection) to Month 1
  Geometric mean titers of neutralizing antibodies against the original strain D614G and the relevant circulating variants measured

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | From Day 0 to the end of the follow-up (Month 6)
  * Proportion of participants with solicited local and systemic Adverse Reactions (ARs): overall; by grade [Time Frame: Up to Day 7 (7 days post vaccination)]
  * Proportion of participants with unsolicited adverse events (AEs): overall; by grade; by relationship to the vaccine [Time Frame: from Day 0 to end of follow-up]
  * Proportion of participants with serious adverse events (SAEs): overall; by grade; by relationship to the vaccine; [Time Frame: from Day 0 to end of follow-up]
Immune response capacity (Immunogenicity) | From Day 0 to Month 6
  * Geometric mean titers and its 95% two-sided confidence interval of neutralizing antibodies against the original strain D614G and the relevant strain circulating.
  * Seroconversion rate and its 95% confidence interval.
  * Geometric mean titers and its 95% confidence interval of IgG binding against the original strain D614G and the relevant circulating variants.
  * Seroconversion rate and its 95% confidence interval.
  * For each relevant VOCs :
    * Geometric mean titers of neutralizing antibodies at Month 1
    * The rate of increase (crude variation of neutralizing antibody titers) between baseline Day0 and Month1and its 95% confidence interval
  * Levels of Cytokine expression patterns of CD4 and CD8 T-cells measured by intracellular cytokine staining assay.
  * Magnitude (percentage) of cells producing at least one cytokine.
  * Spearman correlation coefficient between magnitude of CD4+ specific T-cell responses and humoral responses (titers of neutralizing and IgG binding antibodies, respectively)

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - Centre de Recherche Clinique CHU de Caen Normandie, Caen
  - CIC 1405 CHU Clermont Ferrand, Clermont-Ferrand
  - Hôpital Henri Mondor, Créteil
  - CIC 1403 CHU de Lille, Lille
  - CIC 1413 CHU de Nantes, Nantes
  - CIC 1417 Cochin-Pasteur Hôpital Cochin, Paris
  - CIC 1427 Hôpital St Louis, Paris